CLINICAL TRIAL: NCT06618352
Title: The Effects of Indoor Overheating on Physiological Strain in Young Adults During a Simulated Multi-day Heat Event
Brief Title: Physiological Strain in Young Adults During a Simulated Heat Wave
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Responsible Party: Principal Investigator, Glen P. Kenny, Full Professor, University of Ottawa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HEPRU-2024-09-C
Record Dates: First submitted 2024-09-23; First posted 2024-10-01 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Heat Stress; Physiological Stress
Keywords: Heat wave; Indoor temperatures; Thermoregulation; Heat strain; Young adults; Cardiovascular strain; Sleep; Fatigue
MeSH Terms: conditions — Heat Stress Disorders; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Daylong exposure to extreme heat (Experimental): Young adults exposed to daylong indoor overheating associated with an extreme heat event involving a 10-hour daytime exposure at 36°C (45% relative humidity) followed by a 14-hour nighttime exposure at 31°C (45% relative humidity) over three successive days with only a daytime exposure on the final day.
  Interventions: Other: Simulated indoor overheating exposure

INTERVENTIONS:
Other: Simulated indoor overheating exposure — Young adults exposed to a multi-day extreme heat event

SUMMARY:
The likelihood of exposure to overheated indoor environments is increasing as climate change is exacerbating the frequency and severity of hot weather and extreme heat events. Prolonged exposure to excessive heat stress can result in a deterioration in physiological function leading to a myriad of pathophysiological conditions (e.g., heat exhaustion, acute kidney injury, adverse cardiovascular events, heat stroke) that if left untreated can lead to death. While the relationship between extreme heat events and human health has been assessed in relation to outdoor exposure to high heat conditions, relatively little is known about the effects of daylong exposures to indoor overheating on the body's physiology.

In this study, investigators will examine the change in physiological responses (i.e., thermal, cardiovascular) in young (18-35 years) adults exposed to successive days and nights of high indoor temperatures typical of conditions recording in dwellings without air conditioning during the 2021 Western Heat Dome. Specifically, study participants will be housed in a large environmental chamber (outfitted with bed, work space, sitting area, kitchen and bathroom) for three successive days (three days and two nights) while exposed to indoor overheating where daytime temperatures will be maintained at 36°C (45% relative humidity; note: 36°C, temperatures experienced in homes without air-conditioning) for a 10-hour daytime exposure period (DAYTIME: defined as the time period from 9:00 to 19:00). For the nighttime exposure period (NIGHTTIME: defined as the time period from 19:00 to 9:00), participants will be exposed to nighttime temperatures fixed at 31°C (45% relative humidity; note: reductions in indoor temperatures during the nighttime in large urban centers range between 4-6°C). Participants will be permitted to move freely throughout the day in the chamber, but will be restricted from performing any physical activity except for the completion of a battery of tests (cardiovascular, cognitive and posture assessments performed prior to (as performed between 7:00 and 9:00) and the end (as performed between 17:00 and 19:00) of the daytime exposure). During the nighttime period, participants will be permitted to move freely until they decide to go to bed.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking.
* English or French speaking.
* Ability to provide informed consent.

Exclusion Criteria:

* Chronic health conditions.
* Endurance trained
* Regular exposure to heat (e.g., hot baths, sauna, regular exercise in the heat, recent vacation to area with high temperature).

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-09-28 (Actual); Primary Completion 2025-05-27 (Actual); Study Completion 2025-05-27 (Actual)

PRIMARY OUTCOMES:
Core temperature (Peak) during daytime | End of daytime exposure (hour 10 for Day 1, 2 and 3 of the three day exposure) (daytime defined as period between 9:00 to 19:00)
  Peak rectal temperature (15 min average) during exposure. Rectal temperature is measured continuously throughout the daytime period of the simulated heat wave.
Core temperature (AUC) during daytime | End of daytime exposure (hour 10 for Day 1, 2 and 3 of the three day exposure) (daytime defined as period between 9:00 to 19:00)
  Area under the curve of rectal temperature (in degree-hours)
Core temperature end of daytime exposure | End of daytime exposure (hour 10 for Day 1, 2 and 3 of the three day exposure) (daytime defined as period between 9:00 to 19:00)
  Rectal temperature measured at hour 10 of each daytime exposure to simulated heat wave (15-min average)
Heat rate peak during daytime | End of daytime exposure (hour 10 for Day 1, 2 and 3 of the three day exposure) (daytime defined as period between 9:00 to 19:00)
  Heart rate during each daytime exposure to simulated heat wave (15-min average)
Heat rate AUC during daytime | End of daytime exposure (hour 10 for Day 1, 2 and 3 of the three day exposure) (daytime defined as period between 9:00 to 19:00)
  Heart rate measured during each daytime exposure to simulated heat wave (15-min average)
Cardiac response to standing from supine (30:15 Ratio) during daytime | At the start (hour 0) and end of daytime exposure (hour 10 for Day 1, 2 and 3 of the three day exposure) (daytime defined as period between 9:00 to 19:00)
  Cardiac response to standing evaluated as the ratio between the highest R-wave to R-wave interval (lowest heart rate) measured at the 30th heart beat after standing from supine (+/- 5 beats) and the lowest R-wave to R-wave interval (highest heart rate) measured at the 15th heart beat after standing (+/- 5 beats). Cardiac response to standing will be evaluated twice, during two lying-to-standing tests (separated by 10 min of supine rest). Assessment is perform in the morning prior to ( and following daytime exposure.
Cognitive function during daytime | At the start (hour 0) and end of daytime exposure (hour 10 for Day 1, 2 and 3 of the three day exposure) (daytime defined as period between 9:00 to 19:00)
  Participants will be provided with a tablet device with the mobile testing platform (Sway Medical). Participants will be complete the following cognitive tests below:
  Reaction time: participants will be asked to initiate a movement of the device in response to a visual cue.
  Impulse control: participants will be asked to respond to both "go" and "no-go" visual cues. In response to the "go" cue, participants will initiate a movement of the device.
  Memory: participants complete both a delayed recall test and a working memory test.
  Executive function: participants will complete the Cued Stroop test, in which they are presented a sequence of congruent, neutral and incongruent colour-word tasks.
Postural stability during daytime | At the start (hour 0) and end of daytime exposure (hour 10 for Day 1, 2 and 3 of the three day exposure) (daytime defined as period between 9:00 to 19:00)
  Balance will be assessed in two ways:
  Method 1: CDC 4-Stage Balance Test. Participants hold a tablet to their chest, then auditory cues guide participants through four consecutive stances, feet side by side, instep of one foot touching the big toe of the other foot, tandem stand with one foot in front of the other, heel touching toe, and stand on one foot. The balance assessment will be evaluated based on movement detected by an accelerometer integrated into the hardware of the tablet device (Sway Medical Inc).
  Method 2: Participants will be asked to stand on a BTracks force plate with their feet spread out to shoulder width, hand on their hips and eyes closed. The assessment will comprise of four trials (one practice trial) lasting 20 seconds in length and 20 seconds between trials. Center of pressure (COP) vector data along vertical (y) and horizontal (x) axes will be summed for the total path excursion length (cm) during each trial.
Systolic Response to Standing From Supine during daytime | At the start (hour 0) and end of daytime exposure (hour 10 for Day 1, 2 and 3 of the three day exposure) (daytime defined as period between 9:00 to 19:00)
  Systolic blood pressure response to standing evaluated as the difference in blood pressure measured between the standing and supine. Standing systolic blood pressure will be taken as the lowest value of those measured after 60 and 120 seconds of standing. Systolic response to standing will be evaluated twice, during two lying-to-standing tests (separated by 10 min of supine rest).
Systolic blood pressure during daytime | End of daytime exposure (hour 10 for Day 1, 2 and 3 of the three day exposure) (daytime defined as period between 9:00 to 19:00)
  Systolic blood pressure measured in triplicate via automated oscillometry (~60 seconds between measures)
Diastolic blood pressure during daytime | End of daytime exposure (hour 10 for Day 1, 2 and 3 of the three day exposure) (daytime defined as period between 9:00 to 19:00)
  Diastolic blood pressure measured in triplicate via automated oscillometry (~60 seconds between measures)
Rate pressure product during daytime | End of daytime exposure (hour 10 for Day 1, 2 and 3 of the three day exposure) (daytime defined as period between 9:00 to 19:00)
  Rate pressure product, an index of myocardial work and strain, calculated as systolic blood pressure x heart rate.
Heart rate variability: SDNN during daytime | End of daytime exposure (hour 10 for Day 1, 2 and 3 of the three day exposure) (daytime defined as period between 9:00 to 19:00)
  Standard deviation of normal-to-normal R-wave to R-wave intervals (SDNN) measured during 5 minutes of paced breathing (15 breaths/min) with participants in the seated position. SDNN will be evaluated twice, during two paced breathing periods (separated by 4 min of seated rest).
Heart rate variability: RMSSD during daytime | End of daytime exposure (hour 10 for Day 1, 2 and 3 of the three day exposure) (daytime defined as period between 9:00 to 19:00)
  Root mean squared standard deviation of normal-to-normal R-wave to R-wave intervals (RMSSD) measured during 5 minutes of paced breathing (15 breaths/min) with participants in the seated position. RMSSD will be evaluated twice, during two paced breathing periods (separated by 4 min of seated rest).
Fluid consumption during daytime | End of daytime exposure (hour 10 for Day 1, 2 and 3 of the three day exposure) (daytime defined as period between 9:00 to 19:00)
  Average hourly fluid consumption calculated by weighing participant water intake at the start and end of each hour of exposure (normalized to the exposure duration).
Fluid loss during daytime | End of daytime exposure (hour 10 for Day 1, 2 and 3 of the three day exposure) (daytime defined as period between 9:00 to 19:00)
  Fluid loss calculated as the change in body mass during each exposure presented as a percentage of baseline body mass (corrected for food consumption)
Change in plasma volume during daytime | End of daytime exposure (hour 10 for Day 1, 2 and 3 of the three day exposure) (daytime defined as period between 9:00 to 19:00)
  Change in plasma volume from baseline values calculated from duplicate measurements of hemoglobin and hematocrit at the start and end of each exposure using the technique by Dill and Costill
Thermal comfort scale during daytime | End of daytime exposure (hour 10 for Day 1, 2 and 3 of the three day exposure) (daytime defined as period between 9:00 to 19:00)
  Thermal comfort assessed via a visual analog scale ("How comfortable does your body temperature feel?") ranging from "extremely uncomfortable" to "extremely comfortable"(midpoint: neutral).
Thermal sensation scale during daytime | End of daytime exposure (hour 10 for Day 1, 2 and 3 of the three day exposure) (daytime defined as period between 9:00 to 19:00)
  Thermal sensation assessed via a visual analog scale ("How hot do you feel?") ranging from "extremely hot" to "neutral"(midpoint: hot).
Thirst sensation scale during daytime | End of daytime exposure (hour 10 for Day 1, 2 and 3 of the three day exposure) (daytime defined as period between 9:00 to 19:00)
  Thirst sensation scale assessed via a visual analog scale ("How thirsty are you?") ranging from "Very, very thirsty" to "Not thirsty at all" (midpoint: moderately thirsty).
Arousal scale during daytime | End of daytime exposure (hour 10 for Day 1, 2 and 3 of the three day exposure) (daytime defined as period between 9:00 to 19:00)
  Felt arousal scale assessed via a visual analog scale ("How worked up are you?") ranging from "high arousal" to "low arousal".
Orthostatic intolerance symptoms assessment during daytime | End of daytime exposure (hour 10 for Day 1, 2 and 3 of the three day exposure) (daytime defined as period between 9:00 to 19:00)
  Cumulative sum of scores on 6 questions asking participant to rank symptoms associated with orthostatic intolerance during the lying to standing tests. All symptoms scored on a scale from 0 (none) to 10 (worst possible) and include feelings of: (1) "dizziness, lightheadedness, feeling faint, or feeling like you might black out"; (2) "Problems with vision (blurring, seeing spots, tunnel vision, etc.)"; (3) "Weakness"; (4) "Fatigue"; (5) "Trouble concentrating"; and (6) "Head and neck discomfort".
Core temperature (Peak) during nighttime | End of nighttime exposure (hour 24 for Day 1 and Day 2 of the three day exposure; no nighttime exposure for Day 3) (daytime defined as period between 19:00 to 9:00)
  Peak rectal temperature (15 min average) during exposure. Rectal temperature is measured continuously throughout the daytime period of the simulated heat wave.
Core temperature (AUC) during nighttime | End of nighttime exposure (hour 24 for Day 1 and Day 2 of the three day exposure; no nighttime exposure for Day 3) (daytime defined as period between 19:00 to 9:00)
  Area under the curve of rectal temperature (in degree-hours)
Core temperature end of nighttime | End of nighttime exposure (hour 24 for Day 1 and Day 2 of the three day exposure; no nighttime exposure for Day 3) (daytime defined as period between 19:00 to 9:00)
  Rectal temperature measured at hour 10 of each daytime exposure to simulated heat wave (15-min average)
Heat rate peak during nighttime | End of nighttime exposure (hour 24 for Day 1 and Day 2 of the three day exposure; no nighttime exposure for Day 3) (daytime defined as period between 19:00 to 9:00)
  Heart rate during each daytime exposure to simulated heat wave (15-min average)
Heat rate AUC during nighttime | End of nighttime exposure (hour 24 for Day 1 and Day 2 of the three day exposure; no nighttime exposure for Day 3) (daytime defined as period between 19:00 to 9:00)
  Heart rate measured during each daytime exposure to simulated heat wave (15-min average)
Heart rate variability: SDNN during nighttime | End of nighttime exposure (hour 24 for Day 1 and Day 2 of the three day exposure; no nighttime exposure for Day 3) (daytime defined as period between 19:00 to 9:00)
  Standard deviation of normal-to-normal R-wave to R-wave intervals (SDNN) measured during 5 minutes of paced breathing (15 breaths/min) with participants in the seated position. SDNN will be evaluated twice, during two paced breathing periods (separated by 4 min of seated rest).
Heart rate variability: RMSSD during nighttime | End of nighttime exposure (hour 24 for Day 1 and Day 2 of the three day exposure; no nighttime exposure for Day 3) (daytime defined as period between 19:00 to 9:00)
  Root mean squared standard deviation of normal-to-normal R-wave to R-wave intervals (RMSSD) measured during 5 minutes of paced breathing (15 breaths/min) with participants in the seated position. RMSSD will be evaluated twice, during two paced breathing periods (separated by 4 min of seated rest).

SECONDARY OUTCOMES:
Muscle oxygen during battery of cardiovascular, postural and cognitive tests during daytime | End of daytime exposure (hour 10 for Day 1, 2 and 3 of the three day exposure) (daytime defined as period between 9:00 to 19:00)
  Participants will be attached with 2 probes to measure tissue oxygenation on two locations via a non-invasive tool: near-infrared spectroscopy (NIRS). The device (Portalite, Artinis Medical, The Netherlands) is placed on the left prefrontal cortex and muscle belly of the vastus lateralis. It measures local oxy-, deoxy- and total hemoglobin concentration changes and tissue saturation index (TSI) on the specific location of the human body and provide valuable insights during a diverse set of tests.
Profiles of Mood States (POMS) during daytime | End of daytime exposure (hour 10 for Day 1, 2 and 3 of the three day exposure) (daytime defined as period between 9:00 to 19:00)
  Potential changes in mood (7 subscales of mood: tension, anger, depression, fatigue, confusion, vigor and esteem-related affect). The POMS-40 is a validated, self-administered questionnaire that examines seven distinct aspects of mood state across two positive subscales (Esteem-Related Affect, and Vigor) and five negative subscales (Fatigue, Tension, Confusion, Anger, and Depression), which are described across 40 distinct adjectives (reference). For each individual item, participants were asked to describe "how you feel right now" by responding using a 5-point Likert scale (0 = "Not at all", 1 = "A little", 2 = "Moderately", 3 = "Quite a lot", or 4 = "Extremely"). The values of items associated with a specific subscale (e.g., Fatigue) were summed to calculate its score.
Environmental Symptoms Questionnaire (ESQ) | End of daytime exposure (hour 10 for Day 1, 2 and 3 of the three day exposure) (daytime defined as period between 9:00 to 19:00)
  Self-reported environmental reactions and medical symptomatology associated with prolonged heat exposure. The ESQ-IV is a validated 68-item, self-administered questionnaire that has been used successfully in identifying symptomatology during exposure to a wide variety of environmental conditions, including heat exposure [24, 25]. Participants are asked to assess and described "how you have been feeling today" by responding to each item using a 6-point Likert scale (0 = "Not at all", 1 = "Slight", 2 = "Somewhat", 3 = "Moderate", 4 = "Quite a bit", or 5 = "Extreme"). Total Symptom Score was calculated from this data by taking the sum of the intensity ratings from all 68 individual items using reverse scores for the three positive items from the list ("I Felt Good", "I Felt Alert", and "I Felt Wide Awake").
Sleep quality and quantify assessment | End of daytime exposure (hour 10 for Day 1, 2 and 3 of the three day exposure) (daytime defined as period between 9:00 to 19:00)
  The following questionnaires will be administered:
  * Consensus Sleep Diary (CSD) to provide an overview of the sleep quantity and quality of the previous night.
  * Richards-Campbell Sleep Questionnaire to evaluate the perception of sleep .
  * Leeds Sleep evaluation questionnaire which is 10-item, subjective, questionnaire designed to assess changes in sleep quality over the course of the intervention.
Sleepiness during daytime | End of daytime exposure (hour 10 for Day 1, 2 and 3 of the three day exposure) (daytime defined as period between 9:00 to 19:00)
  The following questionnaires will be administered to evaluate the participants sleepiness during the daytime exposure period:
  * Karolinska sleepiness scale measures the subjective level of sleepiness at a particular time during the day.
  * Stanford sleepiness scale consists of only one item, where participant must identify one of seven statements that best represents their level of perceived sleepiness

CONTACTS AND LOCATIONS:
Overall Officials: Glen P Kenny, PhD, Principal Investigator — University of Ottawa
Locations (1):
- University of Ottawa, Ottawa, Ontario, Canada